CLINICAL TRIAL: NCT03992300
Title: Comparison of Accuracy and Timing Parameter of Digital and Conventional Impression Techniques on Fully Edentulous Jaws: an in Vivo Study
Brief Title: Comparison of Full-arch Implant-supported Frameworks From an Intraoral Scanning or From a Conventional Impression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Miguel Roig Cayón, Professor and Chair Department of Restorative Dentistry, Universitat Internacional de Catalunya
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: REST-ECT-2017-03
Record Dates: First submitted 2019-06-17; First posted 2019-06-20 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-06

CONDITIONS: Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Intervention Model Description: Two frameworks with the same design obtained from two different models (intraoral scanning and conventional impression) are processed and tested in every patient
Who Masked: Outcomes Assessor
Masking Description: The frameworks are marked with a triangle or a circle in the distal aspect of the distal right molar. The outcomes assessor does not now to which group corresponds each framework
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraoral scanning (Experimental): An intraoral scanning is taken. An auxiliary device is used to achieve better accuracy. A zirconia framework is produced
  Interventions: Device: Clinical adjustment
- Conventional scanning (Active Comparator): A conventional elastomeric impression is taken and a zirconia framework is produced
  Interventions: Device: Clinical adjustment

INTERVENTIONS:
Device: Clinical adjustment — Accuracy of the framework is checked in the patient mouth by tactile perception, screwing torque, Sheffield test and radiography.

SUMMARY:
Purpose: To determine if adjustment of full-arch zirconia frameworks processed on a model obtained with an intraoral scanner and an auxiliary device is not inferior to that of identical frameworks obtained from an elastomeric impression.

Materials and methods: Eight consecutive patients ready for a full-arch rehabilitation on already osseointegrated implants were selected. Two sets of impressions were taken, one open tray with polyether and splinted impression copings and a second one with an intraoral scanner. A verification plaster jig was used for the elastomeric impression and a prefabricated auxiliary device was used to adjust the optical intraoral impressions. Two full-zirconia frameworks with the same design were processed and tested on the patient by two independent calibrated operators. Accuracy of both frameworks was measured by calibrated blinded operators, who determined tactile adjustment, Sheffield test, radiographic adjustment, and screwing torque. Overall perception of adjustment was used to determine the better framework to be delivered to the patient.

Hº: Frameworks obtained from an impression taken with an intraoral scanner are not inferior in accuracy to those obtained from a conventional elastomeric impression

DETAILED DESCRIPTION:
Eight consecutive patients ready for a full-arch rehabilitation on previously osseointegrated implants, and who had received an immediately loaded prosthesis, were selected. All implants had multiunit abutments placed on top. Cases from 4 to 6 implants were accepted, either upper or lower arches. Three sets of impressions were taken to each patient:

Conventional impression:

Open tray impression copings were screwed on top of all implants in the arch using a torque wrench set at 10 N/cm. Impression copings were splinted by means of Triad Gel clear resin, with an at least 3mm diameter in the resin connectors. Once the resin was photo-polymerized a cut was done in the centre of each connection with a 0.3 mm bur, to eliminate possible stress in the structure, and then it was splinted again with a drop of Triad Gel in each cut. A polyether impression was taken by means of a perforated plastic tray, and a master model was fabricated following the manufacturer's instructions. A plaster verification jig was fabricated on the model. After one week the patient came to the dental clinic where vertical dimension of occlusion was determined and the plaster key was screwed in the patient mouth to check passivity. In case the key had been fractured, a new impression would have been taken, and if not, final prosthesis could be processed.

Optical impression:

An impression of the antagonist and an impression of the edentulous arch with the healing abutments in place were taken by means of an optical scanner following the manufacturers protocol. The position of the implants was marked in the working standard tessellation language (STL) model, and the software cut a circle on top of those areas. The files were copied, and two datasets were obtained.

Scan-bodies were placed on top of each multiunit abutment, the first STL dataset was open and a second impression was taken, so that the scan-bodies were positioned on the working file.

Scan-bodies were then removed from the patient mouth, and temporary copings were placed on top of each multiunit abutment. A MedicalFit device was selected, and holes were drilled in the position of the implants until it fitted on top of all the cylinders. Cylinders were then splinted to MedicalFit device by means of Triad Gel clear. The device was then removed from the patient mouth and scan implant replicas were placed at the bottom of the metal cylinders. Finally, the device with the scan implant replicas was scanned with an intraoral optical scanner.

The following set of pictures were taken: Rest position, maximum smile (with the scan bodies placed in the mouth), front with retractors (with the scan bodies), and 45º with retractors (also with the scan bodies in place).

All pictures and STL datasets were sent to the dental technician to produce a temporary structure. The STL dataset from the scanning of Medicalfit device used was adjusted to the original STL dataset of the device in the library, and then superimposed to the dataset of the scan-bodies received from us, to allow repositioning of the scan-bodies and to correct possible discrepancies during the intraoral scanning process.

A temporary polymethylmethacrylate (PMMA) framework was delivered by the dental lab and tried in the patient mouth. Corrections were done to adjust occlusion, gingival contour and esthetic parameters where needed. Once esthetic parameters and occlusal scheme were considered correct, a new intraoral scanning was taken with the temporary framework in place. In case changes were done in the gingival contour, scanning of the gingival aspect of the PMMA framework was also done. The PMMA temporary was then left in the patient mouth.

Three pictures were taken with the PMMA framework placed in the mouth: Front full face at rest, front full-face smiling, front full face with separators and full face smiling at 45º.

Clinical adjustment assessment:

After one week two sets of the final prosthesis in full-zirconia were sent from the dental lab, one processed with conventional models and the second fully digital. Both sets were tested in the patient mouth by two calibrated blinded independent operators.

Misfit should be ideally measured in terms smaller than 10 microns, but clinical adjustment is difficult to assess using conventional or quantitative methods. In this research adjustment was assessed following four criteria: passivity in the insertion of the screws, tactile sensation, radiographs and screwing torque:

1. A Visual Analogue Scale (VAS) was used to assess the perception of passivity in the insertion of the prosthodontic screws. A ten centimeters line will be shown to the observer. One side of the line represents "perfect passivity", and the other "no passive at all". The observer will mark his passivity perception on the line between the two endpoints. The distance between "no passivity at all" and the mark will defines the passivity perception.
2. Examination of the marginal fit with an exploratory probe (#23/3 explorer) under 3,8x magnification. Three possible scores were possible: 0 (no gap perceived when probing), 1 (perception of the gap without entering it) and 2 (the tip of the explorer clearly entered the gap).
3. Periapical radiographs were taken with a positioning system to evaluate possible gaps. Five possible scores were possible from 1 to 5, being 1 no gap and increasing 0.15 mm each score until reaching 0.60 mm in score 5.
4. Digital photographs were taken with a 105 mm macro lens. The pictures were calibrated with the known height of the framework and the gap was measured. Four possible scores were possible, being 1 no gap and increasing 0.25 mm each score until reaching 0.75 mm in score 5.
5. Screwing torque on each abutment was measured with the app software from Ichiropro motor (BienAir, Bienne, Switzerland). All screws were hand screwed and then all but the most distal right were unscrewed. Torque was set at 15 N/cm and speed at 5 rpm. The most right distal screw was tightened first, and then the rest of the screws were tightened starting at the most mesial left, following to the most distal left, and from that to the next neighbor implant until all screws were tightened. The torque-time signature was studied in every screw to determine if the torque started to grow just at the end of the tightening or throughout the process. Three scores were possible: 1 for linear value with a fast increase at end of the tightening, 2 for soft continuous growth with a steeper increase at the end, 3 for steep increase at the beginning of tightening.

Once the assessment of the two frameworks was completed, the framework with better adjustment will be placed in the patient, after assessing the presence of correct occlusion, phonetics and esthetic parameters. The second set will be packed and delivered to the patient as a possible replacement in case of problems in the future.

ELIGIBILITY:
Inclusion Criteria:

·Patients with four or more implants already osseo-integrated ready to rehabilitate with a full-arch implant-supported framework of 10 or more units. ·Upper or lower jaw.

Exclusion Criteria:

* Implants not suitable for multiunit abutments.
* More than six implants.
* Peri-implantitis present in any implant.
* Need of a removable prosthesis.
* Patients unable to understand the purpose of the study.
* Patients with a restorative space higher than 15 milimiters.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Accuracy of the framework | one day
  Overall perception of adjustment of the two frameworks

SECONDARY OUTCOMES:
Perception of the passivity | 1 day
  A Visual Analogue Scale (VAS) will be used to assess the perception of passivity in the insertion of the prosthodontic screws. A ten centimeters line will be shown to the observer. One side of the line represents "perfect passivity", and the other "no passivity at all". The observer will mark his passivity perception on the line between the two endpoints. The distance between "no passivity at all" and the mark will define the passivity perception.
Optical adjustment | 1 day
  Examination of the marginal fit with an exploratory probe (#23/3 explorer) under 3,8x magnification. Three possible scores were possible: 0 (no gap perceived when probing), 1 (perception of the gap without entering it) and 2 (the tip of the explorer clearly entered the gap).
Radiographic adjustment | 1 day
  Periapical radiographs will be taken with a positioning system to evaluate possible gaps. Five possible scores will be possible from 1 to 5, being 1 no gap and increasing 0.15mm each score until reaching 0.60mm in score 5.
Screwing torque | 1 day
  Screwing torque in each abutment will be measured by means of Ichiropro® motor. The torque/angle signature will be registered and three possible scores will be possible: 1 for linear value with a fast increase at end of the tightening, 2 for soft continuous growth with a steeper increase at the end, 3 for steep increase at the beginning of tightening.

CONTACTS AND LOCATIONS:
Overall Officials: MIGUEL ROIG CAYON, MD DDS PHD, Study Director — Unversitat Internacional de Catalunya
Locations (1):
- Clinica Universitaria d'Odontologia, Sant Cugat Del Vallés, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
We plan to publish the data in a paper

REFERENCES:
- [Background] Lee H, So JS, Hochstedler JL, Ercoli C. The accuracy of implant impressions: a systematic review. J Prosthet Dent. 2008 Oct;100(4):285-91. doi: 10.1016/S0022-3913(08)60208-5. PMID 18922257
- [Background] al-Turki LE, Chai J, Lautenschlager EP, Hutten MC. Changes in prosthetic screw stability because of misfit of implant-supported prostheses. Int J Prosthodont. 2002 Jan-Feb;15(1):38-42. PMID 11887597
- [Background] Jansen VK, Conrads G, Richter EJ. Microbial leakage and marginal fit of the implant-abutment interface. Int J Oral Maxillofac Implants. 1997 Jul-Aug;12(4):527-40. PMID 9274082
- [Background] Millington ND, Leung T. Inaccurate fit of implant superstructures. Part 1: Stresses generated on the superstructure relative to the size of fit discrepancy. Int J Prosthodont. 1995 Nov-Dec;8(6):511-6. PMID 8595110
- [Background] Sahin S, Cehreli MC. The significance of passive framework fit in implant prosthodontics: current status. Implant Dent. 2001;10(2):85-92. doi: 10.1097/00008505-200104000-00003. PMID 11450418
- [Background] Abduo J, Bennani V, Waddell N, Lyons K, Swain M. Assessing the fit of implant fixed prostheses: a critical review. Int J Oral Maxillofac Implants. 2010 May-Jun;25(3):506-15. PMID 20556249
- [Background] Katsoulis J, Takeichi T, Sol Gaviria A, Peter L, Katsoulis K. Misfit of implant prostheses and its impact on clinical outcomes. Definition, assessment and a systematic review of the literature. Eur J Oral Implantol. 2017;10 Suppl 1:121-138. PMID 28944373
- [Background] Assif D, Marshak B, Schmidt A. Accuracy of implant impression techniques. Int J Oral Maxillofac Implants. 1996 Mar-Apr;11(2):216-22. PMID 8666454
- [Background] Al-Meraikhi H, Yilmaz B, McGlumphy E, Brantley W, Johnston WM. In vitro fit of CAD-CAM complete arch screw-retained titanium and zirconia implant prostheses fabricated on 4 implants. J Prosthet Dent. 2018 Mar;119(3):409-416. doi: 10.1016/j.prosdent.2017.04.023. Epub 2017 Jul 15. PMID 28720339
- [Background] Jemt T. Failures and complications in 391 consecutively inserted fixed prostheses supported by Branemark implants in edentulous jaws: a study of treatment from the time of prosthesis placement to the first annual checkup. Int J Oral Maxillofac Implants. 1991 Fall;6(3):270-6. PMID 1813395
- [Background] Klineberg IJ, Murray GM. Design of superstructures for osseointegrated fixtures. Swed Dent J Suppl. 1985;28:63-9. No abstract available. PMID 3904064
- [Background] Gibbs SB, Versluis A, Tantbirojn D, Ahuja S. Comparison of polymerization shrinkage of pattern resins. J Prosthet Dent. 2014 Aug;112(2):293-8. doi: 10.1016/j.prosdent.2014.02.006. Epub 2014 Apr 14. PMID 24726587
- [Background] Papaspyridakos P, Lal K. Computer-assisted design/computer-assisted manufacturing zirconia implant fixed complete prostheses: clinical results and technical complications up to 4 years of function. Clin Oral Implants Res. 2013 Jun;24(6):659-65. doi: 10.1111/j.1600-0501.2012.02447.x. Epub 2012 Mar 13. PMID 22413889
- [Background] Kan JY, Rungcharassaeng K, Bohsali K, Goodacre CJ, Lang BR. Clinical methods for evaluating implant framework fit. J Prosthet Dent. 1999 Jan;81(1):7-13. doi: 10.1016/s0022-3913(99)70229-5. PMID 9878969
- [Background] Ebadian B, Rismanchian M, Dastgheib B, Bajoghli F. Effect of different impression materials and techniques on the dimensional accuracy of implant definitive casts. Dent Res J (Isfahan). 2015 Mar-Apr;12(2):136-43. PMID 25878678
- [Background] Chochlidakis KM, Papaspyridakos P, Geminiani A, Chen CJ, Feng IJ, Ercoli C. Digital versus conventional impressions for fixed prosthodontics: A systematic review and meta-analysis. J Prosthet Dent. 2016 Aug;116(2):184-190.e12. doi: 10.1016/j.prosdent.2015.12.017. Epub 2016 Mar 2. PMID 26946916
- [Background] Rodriguez JM, Bartlett DW. The dimensional stability of impression materials and its effect on in vitro tooth wear studies. Dent Mater. 2011 Mar;27(3):253-8. doi: 10.1016/j.dental.2010.10.010. Epub 2010 Nov 13. PMID 21075442
- [Background] Thongthammachat S, Moore BK, Barco MT 2nd, Hovijitra S, Brown DT, Andres CJ. Dimensional accuracy of dental casts: influence of tray material, impression material, and time. J Prosthodont. 2002 Jun;11(2):98-108. PMID 12087547
- [Background] Amin WM, Al-Ali MH, Al Tarawneh SK, Taha ST, Saleh MW, Ereifij N. The effects of disinfectants on dimensional accuracy and surface quality of impression materials and gypsum casts. J Clin Med Res. 2009 Jun;1(2):81-9. doi: 10.4021/jocmr2009.04.1235. Epub 2009 Jun 21. PMID 22505972
- [Background] Holst S, Blatz MB, Bergler M, Goellner M, Wichmann M. Influence of impression material and time on the 3-dimensional accuracy of implant impressions. Quintessence Int. 2007 Jan;38(1):67-73. PMID 17216911
- [Background] Schaefer O, Schmidt M, Goebel R, Kuepper H. Qualitative and quantitative three-dimensional accuracy of a single tooth captured by elastomeric impression materials: an in vitro study. J Prosthet Dent. 2012 Sep;108(3):165-72. doi: 10.1016/S0022-3913(12)60141-3. PMID 22944312
- [Background] Zimmermann M, Mehl A, Mormann WH, Reich S. Intraoral scanning systems - a current overview. Int J Comput Dent. 2015;18(2):101-29. English, German. PMID 26110925
- [Background] Menini M, Setti P, Pera F, Pera P, Pesce P. Accuracy of multi-unit implant impression: traditional techniques versus a digital procedure. Clin Oral Investig. 2018 Apr;22(3):1253-1262. doi: 10.1007/s00784-017-2217-9. Epub 2017 Sep 30. PMID 28965251
- [Background] Ahlholm P, Sipila K, Vallittu P, Jakonen M, Kotiranta U. Digital Versus Conventional Impressions in Fixed Prosthodontics: A Review. J Prosthodont. 2018 Jan;27(1):35-41. doi: 10.1111/jopr.12527. Epub 2016 Aug 2. PMID 27483210
- [Background] Tan MY, Yee SHX, Wong KM, Tan YH, Tan KBC. Comparison of Three-Dimensional Accuracy of Digital and Conventional Implant Impressions: Effect of Interimplant Distance in an Edentulous Arch. Int J Oral Maxillofac Implants. 2019 March/April;34(2):366-380. doi: 10.11607/jomi.6855. Epub 2018 Dec 5. PMID 30521661
- [Background] Penarrocha-Diago M, Balaguer-Marti JC, Penarrocha-Oltra D, Balaguer-Martinez JF, Penarrocha-Diago M, Agustin-Panadero R. A combined digital and stereophotogrammetric technique for rehabilitation with immediate loading of complete-arch, implant-supported prostheses: A randomized controlled pilot clinical trial. J Prosthet Dent. 2017 Nov;118(5):596-603. doi: 10.1016/j.prosdent.2016.12.015. Epub 2017 Apr 3. PMID 28385445
- [Background] Pradies G, Ferreiroa A, Ozcan M, Gimenez B, Martinez-Rus F. Using stereophotogrammetric technology for obtaining intraoral digital impressions of implants. J Am Dent Assoc. 2014 Apr;145(4):338-44. doi: 10.14219/jada.2013.45. PMID 24686966
- [Background] Corominas-Delgado C, Espona J, Lorente-Gascon M, Real-Voltas F, Roig M, Costa-Palau S. Digital implant impressions by cone-beam computerized tomography: a pilot study. Clin Oral Implants Res. 2016 Nov;27(11):1407-1413. doi: 10.1111/clr.12754. Epub 2015 Dec 30. PMID 26715129
- [Background] Ercoli C, Geminiani A, Feng C, Lee H. The influence of verification jig on framework fit for nonsegmented fixed implant-supported complete denture. Clin Implant Dent Relat Res. 2012 May;14 Suppl 1:e188-95. doi: 10.1111/j.1708-8208.2011.00425.x. Epub 2011 Dec 16. PMID 22176765
- [Background] Alhashim A, Flinton RJ. Dental gypsum verification jig to verify implant positions: a clinical report. J Oral Implantol. 2014 Aug;40(4):495-9. doi: 10.1563/AAID-JOI-D-12-00196. No abstract available. PMID 25106015
- [Background] Jemt T, Rubenstein JE, Carlsson L, Lang BR. Measuring fit at the implant prosthodontic interface. J Prosthet Dent. 1996 Mar;75(3):314-25. doi: 10.1016/s0022-3913(96)90491-6. PMID 8648581